CLINICAL TRIAL: NCT05249751
Title: Copeptin; A Neuroendocrine Biomarker of COVID-19 Severity
Brief Title: Copeptin in COVID-19
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Elshafei, Professor Assistant of Medical Biochemistry and Molecular Biology, Al-Azhar University
Other Study IDs: Al-Azhar Pharmacy
Record Dates: First submitted 2022-02-18; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild-moderate: Cases classified as mild-moderate fulfilled the following criteria: fever and respiratory symptoms, CORAD 1-5, and oxygen saturation (SpO2 92 percent),
  Interventions: Diagnostic Test: Assessement of serum copeptin by ELISA technique
- Severe: severe cases met the following criteria: fever and respiratory symptoms, CORAD 4-5, and oxygen saturation (SpO2 92 percent).
  Interventions: Diagnostic Test: Assessement of serum copeptin by ELISA technique

INTERVENTIONS:
Diagnostic Test: Assessement of serum copeptin by ELISA technique — Assessement of serum copeptin by ELISA technique

SUMMARY:
This study aimed to investigate the change in serum level of copeptin, a neuroendocrine biomarker, in differentiation between mild-moderate and severe COVID-19 cases on admission time and to find its diagnostic potential.

DETAILED DESCRIPTION:
This prospective study enrolled 160 individuals with confirmed COVID-19 infection using PCR. They were recruited from Al-Zahraa Hospital, Faculty of Medicine (Girls), Al-Azhar University, Cairo, Egypt, which was specifically designated for the isolation of SARS-CoV-2 positive patients. According to the Egyptian ministry of health and population's (MOHP) recommendations, patients were divided into 80 mild-moderate COVID-19 patients and 80 severe COVID-19 patients. Cases classified as mild-moderate fulfilled the following criteria: fever and respiratory symptoms, CORAD 1-5, and oxygen saturation (SpO2 92 percent), while severe cases met the following criteria: fever and respiratory symptoms, CORAD 4-5, and oxygen saturation (SpO2 92 percent). All participants or their corresponding companions signed a free informed consent form. The study was approved by the research ethics committee of Al-Azhar University's Faculty of Medicine (Girls), Cairo, Egypt, with approval number (202106884), and adhered to the Helsinki Declaration's precepts. Pregnancy, COVID-19 patients with morbid obesity, cancer, or autoimmune disease, and those who took immunomodulators or initiated the COVID-19 treatment programme were excluded. Additionally, patients having a history of recurrent COVID-19 infection were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

Adult patients > 18 years with the positive result of real-time reverse transcriptase-polymerase chain reaction assay (RT-PCR) for SARS-CoV-2 RNA.

Severity stratification is based on the guidance of the Egyptian MOH protocol.

Exclusion Criteria:

Pregnant COVID-19 patients. COVID-19 patients with morbid obesity, malignancy, autoimmune diseases and those who received immunomodulators or began COVID-19 treatment protocol.

Also, patients with a history of recurrent COVID-19 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian patients recruited from Al-Zahraa Hospital, Faculty of Medicine (Girls), Al-Azhar University, Cairo, Egypt
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
The role of Copeptin in severity stratification of CoVID-19 | By the end of the study (September 2021)
  to determine the effect of COVID-19 severity on the serum copeptin level, which serves as a stress indicator for infection-related complications. Additionally, to link this effect with that of COVID-19's other inflammatory biomarkers, including C-reactive protein (CRP), ferritin, and D-dimer. Additionally, to investigate its utility as a differentiating factor amongst COVID-19 severity classes.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahraa Hospital, Al-Azhar University, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Through the published research article